CLINICAL TRIAL: NCT07288125
Title: The Effect of Cold Atmospheric Plasma on Patient Comfort During Dental Infiltration Anesthesia: A Randomized Controlled Split-Mouth Clinical Trial
Brief Title: Effect of Cold Atmospheric Plasma on Patient Comfort During Dental Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Izzet Acikan, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Harran university HRÜ/25.13.39
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cold Atmospheric Plasma; Dental Anesthesia
Keywords: Cold Atmospheric Plasma; Local Anesthesia; Injection Pain; Dental Anxiety
MeSH Terms: interventions — Plasma Gases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP (Experimental): Cold Atmospheric Plasma applied before injection
  Interventions: Other: Cold Atmospheric Plasma
- Control (Active Comparator): No pretreatment, standard injection only
  Interventions: Other: No pretreatment

INTERVENTIONS:
Other: Cold Atmospheric Plasma — Cold atmospheric plasma is applied to the oral mucosa at the planned injection site for 30 seconds using a non-contact atmospheric plasma device before local infiltration anesthesia.
  Arms: CAP
Other: No pretreatment — No pretreatment is applied. The control side receives only the standard buccal local infiltration anesthesia.
  Arms: Control

SUMMARY:
This study aims to investigate the effectiveness of cold atmospheric plasma, a laser-like biophysical method, in reducing injection pain experienced during local infiltration anesthesia in dental treatments. The purpose is to determine whether applying cold atmospheric plasma before the injection can decrease the level of pain at the injection site and improve patient comfort.

In this study, to help reduce the pain felt during the dental injection, some patients will receive a cold plasma application before the needle is administered. The device is held close to the gum area where the injection will be given-without touching the tissue-for about one minute to help the area relax. Afterwards, the standard local anesthetic injection is performed. On the opposite side of the mouth, only the normal injection will be given. Pain levels on both sides and patient satisfaction will be recorded through questions asked after the procedure.

If you choose to participate in this research, your dental treatments will still be completed, and the pain felt during the injection may be reduced. Additionally, by participating, you will contribute to scientific knowledge and to the development of a potential future treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years of age;
* American Society of Anesthesiologists (ASA) physical status classification I (systemically healthy);
* No known allergy or intolerance to local anesthetic agents or cold atmospheric plasma (CAP);
* Presence of similar bilateral dental treatment indications in the maxilla or mandible.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Presence of active lesions, ulceration, or signs of infection in the mucosa at the injection site;
* Immunodeficiency or systemic immunosuppressive therapy;
* Use of anticoagulant medications;
* Previous exposure to CAP therapy for any purpose;
* History of allergy to local anesthetic agents;
* Presence of neurological or psychiatric disorders that may affect pain perception.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity During Local Anesthesia Injection | Immediately after injection
  The primary outcome was the intensity of pain experienced during the injection, assessed by the patient using a visual analog scale (VAS). The VAS ranged from 0 to 10, where 0 represented "no pain" and 10 represented "unbearable pain." Immediately after

SECONDARY OUTCOMES:
Patient satisfaction related to the injection experience | Immediately after injection
  Patient satisfaction will be assessed using a 15-item Likert-type questionnaire completed after both local anesthesia injections. Each item is scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Patients will rate their experiences for the CAP-treated side and the control side separately. The questionnaire includes both negative statements (e.g., insufficient information, fear of the device/procedure, perceived pain, negative emotions, unwillingness to repeat or recommend the procedure) and positive statements (e.g., adequate information, reduced fear, willingness to accept the method even with additional cost, increased motivation to continue treatment, overall satisfaction). Scores will be used to generate satisfaction profiles for each side.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Faculty of Dentistry, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jagtap B, Bhate K, Magoo S, S N S, Gajendragadkar KS, Joshi S. Painless injections-a possibility with low level laser therapy. J Dent Anesth Pain Med. 2019 Jun;19(3):159-165. doi: 10.17245/jdapm.2019.19.3.159. Epub 2019 Jun 30. PMID 31338422
- [Result] Ucar G, Sermet Elbay U, Elbay M. Effects of low level laser therapy on injection pain and anesthesia efficacy during local anesthesia in children: A randomized clinical trial. Int J Paediatr Dent. 2022 Jul;32(4):576-584. doi: 10.1111/ipd.12936. Epub 2022 Feb 8. PMID 34738278